CLINICAL TRIAL: NCT05794906
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study of Darolutamide Plus Androgen Deprivation Therapy (ADT) Compared With Placebo Plus ADT in Patients With High-risk Biochemical Recurrence (BCR) of Prostate Cancer
Brief Title: A Study to Compare Darolutamide Given With Androgen Deprivation Therapy (ADT) With ADT in Men With Hormone Sensitive Prostate Cancer and Raise of Prostate Specific Antigen (PSA) Levels After Local Therapies
Acronym: ARASTEP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21492; 2022-501343-33-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Biochemically Recurrent Prostate Cancer
Keywords: darolutamide; high risk BCR; PSMA PET imaging
MeSH Terms: interventions — darolutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darolutamide+ADT (Experimental): Participants will receive darolutamide plus ADT twice daily with food for a pre-specified duration of 24 months.
  Interventions: Drug: Darolutamide (BAY1841788, Nubeqa); Other: ADT
- Placebo+ADT (Placebo Comparator): Participants will receive Placebo plus ADT twice daily with food for a pre-specified duration of 24 months.
  Interventions: Other: Placebo matching darolutamide; Other: ADT

INTERVENTIONS:
Drug: Darolutamide (BAY1841788, Nubeqa) — Coated tablet, 300 mg / tablet, oral.
  Arms: Darolutamide+ADT
Other: Placebo matching darolutamide — Coated tablet, oral
  Arms: Placebo+ADT
Other: ADT — Luteinizing hormone-releasing hormone [LHRH] agonist/antagonists

SUMMARY:
Researchers are looking for a better way to treat men at high-risk of biochemical recurrence (BCR) of prostate cancer.

BCR means that in men who had prostate cancer and were treated by either surgery and/ or radiation therapy, the blood level of a specific protein called PSA rises. PSA is a marker of prostate cancer cells activity. The PSA increase means that the cancer has come back even though conventional imaging such as computed tomography (CT) scans, magnetic resonance imaging (MRI) and bone scans does not show any lesion of prostate cancer. Recently a more sensitive imaging method called prostate-specific membrane antigen [PSMA] positron emission tomography [PET]) /computed tomography [CT]) scan may identify prostate cancer lesions not detectable by conventional imaging. Men with BCR have a higher risk of their cancer spreading to other parts of the body, particularly when PSA levels raised to a certain limit within a short period of time after local therapies. Once the cancer spreads to other parts of the body, it can become even harder to treat.

In men with prostate cancer, male sex hormones (also called androgens) like testosterone can help the cancer grow and spread. To reduce androgens levels in these patients, there are treatments that block androgens production in the body called androgen deprivation therapy (ADT). ADT is often used to stop prostate cancer. Another way to stop prostate cancer growth and spread is to block the action of androgen receptors on prostate cancer cells called androgen receptor inhibitors (ARIs). The new generation ARIs including darolutamide can block the action of androgens receptors and are available for the treatment of prostate cancer in addition to ADT. It is already known that men with prostate cancer benefit from these treatments.

The main objective of this study is to learn if the combination of darolutamide and ADT prolongs the time that the participants live without their cancer getting worse, or to death due to any cause, compared to placebo (which is a treatment that looks like a medicine but does not have any medicine in it) and ADT given for a pre-specified duration of 24 months.

To do this, the study team will measure the time from the date of treatment allocation to the finding of new cancer spread in the participants by using PSMA PET/CT, or death due to any cause. The PSMA PET/CT scans is performed using a radioactive substance called a "tracer" that specifically binds to the prostate-specific membrane antigen (PSMA) which is a protein often found in large amounts on prostate cancer cells.

To avoid bias in treatment, the study participants will be randomly (by chance) allocated to one of two treatment groups. Based on the allocated treatment group, the participants will either take darolutamide plus ADT or placebo plus ADT twice daily as tablets by mouth. The study will consist of a test (screening) phase, a treatment phase and a follow-up phase. The treatment duration is pre-specified to be 24 months unless the cancer gets worse, the participants have medical problems, or they leave the study for any reason. In addition, image guided radiotherapy (IGRT) or surgery is allowed and your doctor will explain the benefits and risks of this type of therapy.

During the study, the study team will:

* take blood and urine samples.
* measure PSA and testosterone levels in the blood samples
* do physical examinations
* check the participants' overall health
* examine heart health using electrocardiogram (ECG)
* check vital signs
* check cancer status using PSMA PET/CT scans, CT, MRI and bone scans
* take tumor samples (if required)
* ask the participants if they have medical problems

About 30 days after the participants have taken their last treatment, the study doctors and their team will check the participants' health and if their cancer worsened. The study team will continue to check this and regularly ask the participants questions about medical problems and subsequent therapies until they leave the study for any reason or until they leave the study for any reason or until the end of the study, whatever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent as described which includes compliance with the requirements, restrictions listed in the informed consent form (ICF), and in this protocol.
* Male ≥18 years of age at the time of signing the informed consent.
* Histologically or cytologically confirmed adenocarcinoma of prostate.
* Prostate cancer initially treated by: radical prostatectomy (RP) followed by adjuvant radiotherapy (ART), or salvage radiotherapy (SRT), or RP in participants who are unfit for (or refused) ART or SRT, or primary radiotherapy (RT).
* High-risk biochemical recurrence (BCR), defined as Prostate-specific antigen doubling time (PSADT) <12 months calculated using the formula provided by the Sponsor, and PSA ≥0.2 ng/mL after ART or SRT post RP or after RP in participants who are unfit for ART or SRT (local or central values accepted), or PSA ≥2 ng/mL above the nadir after primary RT only (local or central values accepted).
* Participants must undergo prostate-specific membrane antigen positron emission tomography/computed tomography (PSMA PET/CT) within the 42-day Screening period using either 18F-DCFPyL (piflufolastat F 18) or 68Ga-PSMA-11 which will be assessed by blinded independent central review (BICR) to identify at least one PSMA PET/CT lesion of prostate cancer.
* Serum testosterone ≥150 ng/dL (5.2 nmol/L) (local assessment is allowed whenever central assessment cannot be done).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Blood counts at screening: Hemoglobin ≥9.0 g/dL (participant must not have received blood transfusion within 7 days prior to sample being taken); Absolute neutrophil count (ANC) ≥1.5x10^9/L (participant must not have received any growth factor within 4 weeks prior to sample being taken); Platelet count ≥100x10^9/L.
* Screening values of: Alanine aminotransferase (ALT) ≤1.5 x upper limit of normal (ULN); Aspartate aminotransferase (AST) ≤1.5 x ULN; Total bilirubin (TBL) ≤1.5 ULN, (except participants with a diagnosis of Gilbert's disease); Estimated glomerular filtration rate (eGFR) >40 ml/min/1.73 m^2 calculated by the CKD-EPI formula.
* Sexually active male participants must agree to use contraception as detailed in the protocol during the Treatment period and for at least 1 week after the last dose of study treatment, and refrain from donating sperm during this period.

Exclusion Criteria:

* Pathological finding consistent with small cell, ductal or ≥50 % component of neuroendocrine carcinoma of the prostate.
* History of bilateral orchiectomy.
* Metastases or recurrent /new malignant lesions in prostate gland/bed seminal vesicles, lymph nodes below the CIA bifurcation on conventional imaging (CI) as assessed by BICR during screening.
* Brain metastasis on PSMA PET /CT by BICR at screening.
* High-risk BCR after primary radiotherapy with new loco-regional lesions on screening PSMA PET/CT who are eligible for curative salvage prostatectomy.

Note: Participants treated with curative salvage prostatectomy after primary RT who meet the PSA criteria (inclusion criteria 5) may be considered for the study.

* Prior treatment with second generation (e.g. enzalutamide, apalutamide) androgen receptor inhibitors (ARIs) and CYP 17 inhibitors (e.g., abiraterone) within 18 months prior to signing of the ICF.
* Prior treatments with PSMA-radiotherapeutics within 12 months prior to randomization.
* Prior radiotherapy (including image-guided radiotherapy) as primary, adjuvant or salvage treatment completed within 8 weeks prior to signing of the ICF.
* Any prior malignancy (other than adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) within 5 years.
* History of pelvic radiotherapy for other malignancy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 981 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2030-03-29 (Estimated)

PRIMARY OUTCOMES:
Radiological progression-free survival (rPFS) by Prostate-specific membrane antigen (PSMA) positron emission tomography/computed tomography (PET/CT) assessed by Blinded independent central review (BICR) | After randomization to after last treatment, approximately 24 months

SECONDARY OUTCOMES:
Metastasis-free survival (MFS) by Conventional imaging (CI) assessed by BICR | After randomization to after last treatment, approximately 46 months
Time to Castration-resistant prostate cancer (CRPC) | After randomization to after last treatment, approximately 46 months
Time to initiation of first subsequent systemic antineoplastic therapy | After randomization to after last treatment, approximately 46 months
Time to loco-regional progression by PSMA PET/CT | After randomization to after last treatment, approximately 46 months
Time to first Symptomatic skeletal event (SSE) | After randomization to after last treatment, approximately 46 months
Overall survival (OS) | After randomization to after last treatment, approximately 46 months
Prostate-specific antigen (PSA) undetectable rates (<0.2 ng/mL) | After randomization to after last treatment, approximately 46 months
Time to deterioration in the Functional Assessment of Cancer Therapy-Prostate (FACT-P) total score | After randomization to after last treatment, approximately 24 months
  FACT-P is a multidimension, selfreport QoL instrument specifically designed for patients with prostate cancer. It consists of 39 questions items, made up by 2 parts: the 27 questions for functional assessment of cancer therapy general (FACT-G) and 12 prostate cancer subscale questions. It assesses 4 main domains which are: physical (n=7), social/family (n=7), emotional (n=6) and functional wellbeing (n=7).
Time to symptomatic progression | After randomization to after last treatment, approximately 46 months
Number of participants with Treatment-emergent adverse events (TEAEs) and Treatment-emergent serious adverse events (TESAEs) categorized by severity | After the first treatment until 30 days (+7 days) after the last treatment, up to 25 months
Number of participants who discontinue study treatment due to a TEAE | After the first treatment until 30 days (+7 days) after the last treatment, up to 25 months

CONTACTS AND LOCATIONS:
Locations (228):
- United States (25):
  - Mayo Clinic Hospital - Phoenix - Cardiology, Phoenix, Arizona
  - City of Hope - Duarte Cancer Center, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - UCLA Clark Urology Center, Los Angeles, California
  - UCSF Bakar Precision Cancer Medicine Building - Genitourinary, San Francisco, California
  - Colorado Urology - St. Anthony Hospital Campus, Lakewood, Colorado
  - Northwestern Medicine - Urology, Chicago, Illinois
  - The University of Kansas Cancer Center - Richard and Annette Bloch Radiation Oncology Pavilion, Kansas City, Kansas
  - Chesapeake Urology Associates - Towson, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center - Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute - Oncology Department, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute - Detroit Headquarters, Detroit, Michigan
  - M Health Fairview Masonic Cancer Clinic - Clinics and Surgery Center, Minneapolis, Minnesota
  - Washington University School of Medicine - Center for Advanced Medicine (CAM), St Louis, Missouri
  - XCancer Omaha, Omaha, Nebraska
  - NYU Langone Health, Mineola, New York
  - Icahn School of Medicine at Mount Sinai - Oncology, New York, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Carolina Urological Research Center, Myrtle Beach, South Carolina
  - University Hospital Simmons Cancer Center Genitourinary Clinic, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
  - USA Clinical Trials, San Antonio, Texas
  - The Urology Place, San Antonio, Texas
- Australia (11):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - University of New South Wales (UNSW) - Liverpool Hospital - Liverpool Cancer Therapy Centre, Liverpool, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Clinical Research Unit - Box Hill, Box Hill, Victoria
  - Epworth HealthCare, East Melbourne, Victoria
  - Northern Hospital, Epping, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Western Urology, Maribyrnong, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (6):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Krankenhaus der Barmherzigen Brüder, Vienna, Vienna
  - Medizinische Universitaet Graz - Klinische Abteilung für Onkologie - Innere Medizin, Graz
  - Uniklinikum Salzburg - Landeskrankenhaus, Salzburg
  - Medizinische Universität Wien- Universitätsklinik für Urologie, Vienna
- Belgium (6):
  - Maria Middelares General Hospital | Medical Oncology Department, Ghent
  - UZ Gent - department Urology, Ghent
  - Jessa Hospital | Campus Virga Jesse - Data Management Oncology and Hematology Department, Hasselt
  - AZ Groeninge Campus Kennedylaan - Urology, Kortrijk
  - Hopital de La Louvière - Site Jolimont - Oncology department, La Louvière
  - Universitair Ziekenhuis Leuven | Gasthuisberg Campus - Urology Department, Leuven
- Brazil (18):
  - Oncocentro - Fortaleza, Fortaleza, Ceará
  - Hospital Evangélico de Cachoeiro de Itapemirim, Vitória, Espírito Santo
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Assistência Multidisciplinar em Oncologia (AMO), Salvador, Estado de Bahia
  - Liga Paranaense de Combate ao Cancer-Hosp Erasto Gaertner, Curitiba, Paraná
  - Instituto D'Or Pesquisa e Ensino (IDOR) (D'Or Institute for Research & Education) - Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense Contra o Cancer | Centro de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital Moinhos de Vento-Centro Clínico, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo, São Paulo
  - Inst. de Assistência Médica ao Sérvidor Público Estadual, São Paulo, São Paulo
  - Hospital das Clínicas da Universidade de Campinas - UNICAMP, São Paulo, São Paulo
  - Universidade Estadual do Rio de Janeiro, Rio de Janeiro
  - Hospital Sirio Libanes, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital do Cancer de Sao Paulo - A. C. Camargo, São Paulo
- Canada (16):
  - Prostate Cancer Centre, Calgary, Alberta
  - Kaye Edmonton Clinic - Dianne and Irving Kipnes Urology Centre, Edmonton, Alberta
  - BC Cancer - Abbotsford, Abbotsford, British Columbia
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - St. Joseph's Healthcare - Hamilton, Hamilton, Ontario
  - London Health Sciences Centre (LHSC) - London Regional Cancer Program (LRCP), London, Ontario
  - Princess Margaret Cancer Centre - Oncology Department, Toronto, Ontario
  - Hôtel-Dieu de Lévis - Urology, Québec, Province
  - CISSS de l'Outaouais - Hopital de Gatineau - Centre de cancerolgie, Gatineau, Quebec
  - Urology South Shore Research - Research Department, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital - Radiation Oncology, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS) - Hopital Fleurimont, Sherbrooke, Quebec
  - Centre integre universitaire de sante et de services sociaux de la Mauricie-et-du-Centre-du-Quebec - Radio-oncologie, Trois-Rivières, Quebec
- China (10):
  - Peking University First Hospital - Oncology Department, Beijing, Beijing Municipality
  - Zhongnan hospital ,Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital - Oncology Department, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center - Oncology Department, Shanghai, Jiangsu
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - The 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital (PUMCH) - East Location, Beijing
  - Jiangsu Provincial People's Hospital - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Tianjin Cancer Hospital, Airport Hospital, Tianjin
- Czechia (6):
  - Fakultni nemocnice u Sv. Anny, Onkologicko-chirurgicke oddeleni, Brno
  - Masarykova Univerzita - Masarykuv Onkologicky Ustav (MOU) - Klinika Komplexni Onkologicke Pece (KKOP), Brno
  - Fakultní nemocnice Olomouc - Onkologická klinika, Olomouc
  - Všeobecná fakultní nemocnice v Praze - Urologická klinika, Prague
  - Thomayerova Nemocnice (TN) (Thomayers Hospital) - Onkologicka Klinika 1. LF UK A TN, Prague
  - Fakultní nemocnice Motol a Homolka, Pracovište MOTOL - Onkologická klinika 2. LF UK a FNMH, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet - Kræftbehandling, København Ø
  - Sjællands University hospital Næstved, Næstved
- Finland (4):
  - HUS-Yhtymä, Helsingin yliopistollinen sairaala (HUS) - Urologia, Helsinki, Uusimaa
  - Oulu University Hospital, Oulun yliopistollinen sairaala (OYS), Oulu
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS), Tampere
  - Turku University Hospital, Turun yliopistollinen sairaala (TYKS) - Urologia, Turku
- France (23):
  - Center Hospitalier Michallon - Grenoble - Service d Urologie et de la transplantation Renale, La Tronche, Grenoble Cedex 9
  - Centre d' Oncologie du Pays Basque Clinique Belharra - Bayonne - Oncologie medicale, Bayonne
  - CHRU Besancon - Hopital Jean Minjoz, Besançon
  - CHU Bordeaux - Hopital Pellegrin - Service urologie, Bordeaux
  - Hopital La Cavale Blanche - CHU de Brest - institut de cancerologie et d'imagerie, Brest
  - Centre Hospitalier Universitaire de Clermont Ferrand - Gabriel Montpied - Service Urologie, Clermont-Ferrand
  - APHP - Hopital Henri Mondor - Departement Urologie, Créteil
  - Institut de cancerologie de Bourgogne - Departement radiotherapie, Dijon
  - Centre Georges Francois Leclerc Dijon - service de radiotherapie, Dijon
  - Hopital Claude Huriez - Lille - Urologie, Lille
  - Hopital Prive Le Bois - Centre Bourgogne - Service radiotherapie oncologie, Lille
  - UNICANCER - Centre Leon-Berard (CLB) - Medical oncology, Lyon
  - AP-HM - Hopital de la Timone, Marseille
  - Clinique Clementville, Montpellier
  - HCL - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancerologie Jean Godinot - Departement oncologie medicale, Reims
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Institut Curie - Saint-Cloud, Saint-Cloud
  - Institut de Cancerologie de l'Ouest - Saint Herblain - Unite de therapie precoce, Saint-Herblain
  - ICANS - Institut de Cancerologie de Strasbourg Europe, Strasbourg
  - Institut Claudius Regaud - iUCT Oncopole - Service oncologie, Toulouse
  - Institut de Cancérologie de Lorraine - Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy - Departement Oncologie-Radiotherapie, Villejuif
- Germany (20):
  - Klinikum Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Klinikum der Universität Würzburg, Würzburg, Bavaria
  - Universitätsklinikum der Johann Wolfgang Goethe Universität, Frankfurt am Main, Hesse
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig, Lower Saxony
  - Universitätsmedizin der Georg-August-Universität Göttingen, Göttingen, Lower Saxony
  - Urologicum Duisburg, Duisburg, North Rhine-Westphalia
  - Marienhospital Herne Universitätsklinik, Herne, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony
  - Medizinische Fakultät der Otto-von-Guericke Universität, Magdeburg, Saxony-Anhalt
  - Universitätsklinikum Aachen / Klinik und Poliklinik für Urologie und Kinderurologie, Aachen
  - Marien-Krankenhaus Bergisch Gladbach, Bergisch Gladbach
  - Vivantes Klinikum Am Urban, Berlin
  - Universitätsklinikum Hamburg-Eppendorf - Martini-Klinik am UKE GmbH, Hamburg
  - Universitaetsklinikum Jena - Klinik fuer Urologie, Jena
  - Universitätsklinikum Schleswig-Holstein/ Klinik für Urologie, Kiel
  - Johannes Gutenberg-Universität Mainz - Urologie, Mainz
  - Klinikum Stuttgart / Klinik für Urologie und Transplantationschirurgie, Stuttgart
  - Urologische Gemeinschaftspraxis Wesel, Wesel
- Hungary (6):
  - Semmelweis Egyetem, Altalanos Orvostudomanyi Kar, Urologiai Klinika, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Budapesti Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaz, Nyíregyháza
- Italy (20):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti_Foggia - Oncologia Medica e Terapia Biomolecolare Universitaria, Foggia, Apulia
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale - S. C. Oncologia Clinica Sperimentale Uro-Ginecologica, Napoli, Campania
  - Azienda Unita Sanitaria Locale Di Bologna_Ospedale Bellaria - Oncologia Medica, Bologna, Emilia-Romagma
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Urologia, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria di Modena_Policlinico - Oncologia, Modena, Emilia-Romagna
  - Azienda USL IRCCS di Reggio Emilia_Arcispedale Santa Maria Nuova - S.C. Oncologia Provinciale, Reggio Emilia, Emilia-Romagna
  - Centro di Riferimento Oncologico di Aviano - Oncologia Radioterapica, Aviano, Friuli Venezia Giulia
  - I.F.O. Istituti Fisioterapici Ospitalieri_Ospedale Regina Elena - Urologia, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Degenza di Radioterapia Oncologica, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino - Oncologia Medica 1, Genoa, Liguria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - Oncologia, Bergamo, Lombardy
  - Ospedale San Raffaele s.r.l - Urologia, Milan, Lombardy
  - Humanitas Mirasole S.p.A. - Oncologia Medica ed Ematologia, Rozzano, Lombardy
  - A.O.U. Città della Salute e della Scienza di Torino_Molinette - Urologia U, Turin, Piedmont
  - Azienda Provinciale Per I Servizi Sanitari_Ospedale Santa Chiara - UO Oncologia Medica, Trento, Trentino-Alto Adige
  - A.O. di Perugia_Hospital Santa Maria della Misericordia - S.C. Radioterapia Oncologica, Perugia, Umbria
  - Istituto Oncologico Veneto_Castelfranco Veneto - UOC Urologia Oncologica, Castelfranco Veneto, Veneto
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata - UOC Radioterapia, Roma, Veneto
  - Cliniche Gavazzeni S.p.A - Dipartimento Area Chirurgia Unità Operativa di Urologia, Bergamo
  - Azienda Ospedaliera Santa Croce e Carle - Oncologia, Cuneo
- Japan (6):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - The University of Osaka Hospital, Suita, Osaka
  - Institute of Science Tokyo Hospital, Bunkyo-ku, Tokyo
  - Kyoto University Hospital, Kyoto
- Netherlands (6):
  - Albert Schweitzer Hospital | Internal Medicine - Oncology Department, Dordrecht
  - University Medical Center Groningen | Urology Department, Groningen
  - Tergooi MC | Hilversum - Wetenschapsbureau, Hilversum
  - St. Antonius Ziekenhuis | Utrecht - R&D Interne Geneeskunde, Nieuwegein
  - St. Franciscus Gasthuis, Rotterdam
  - HagaZiekenhuis van Den Haag, The Hague
- New Zealand (4):
  - Canterbury Urology Research Trust, Christchurch, Canterbury
  - Auckland City Hospital, Auckland
  - Tauranga Urology Research Limited, Tauranga
  - MidCentral District Health Board (MDHB) - Palmerston North Hospital (PNH), TBC
- Poland (6):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz
  - Swietokrzyskie Centrum Onkologii, Kielce
  - Centrum Medyczne iMed24, Krakow
  - Medrise Sp. z o.o. Centrum Badan Klinicznych, Lublin
  - Szpital Grochowski im. dr.med. Rafala Masztaka, Warsaw
  - EMC Instytut Medyczny SA - Penta Hospitals Przychodnie, Wroclaw Wejherowska, Wroclaw
- Portugal (5):
  - Instituto Portugues de Oncologia de Lisboa | Unidade de Investigacao Clinica - Departamento de Urologia, Lisbon, Lisbon District
  - Unidade Local Saúde Coimbra, E.P.E, Coimbra
  - Companhia Uniao Fabril | Hospital CUF Tejo - Academic Center - Research Center, Lisbon
  - Luz Saude | Hospital da Luz Lisboa - Centro de Investigacao Clinica, Lisbon
  - Hospital Santa Maria | Centro de Investigacao Clinica, Lisbon
- Spain (15):
  - Complexo Hospitalario Universitario De Santiago | Oncologia Radioterapica, Santiago de Compostela, A Coruña
  - Hospital Universitario Marques De Valdecilla - Urologia, Santander, Cantabria
  - Hospital del Mar I Urologia, Barcelona
  - Fundacio Puigvert | Urologia, Barcelona
  - Hospital Universitari Vall D Hebron | Oncologia Radioterapica, Barcelona
  - Hospital Clinic De Barcelona | Urologia, Barcelona
  - Hospital Universitario Puerta Del Mar | Urologia, Cadiz
  - MD Anderson Cancer Center | Oncologia Radioterapica, Madrid
  - Hospital Universitario Ramon Y Cajal | Oncologia Radioterapica, Madrid
  - Hospital Universitario Hm Sanchinarro | Oncologia, Madrid
  - Hospital Universitario Virgen De La Victoria | Urologia, Málaga
  - Hospital General Universitario Morales Meseguer | Urologia, Murcia
  - Hospital Universitario Virgen Del Rocio S.L. | Urologia, Seville
  - Fundacion Instituto Valenciano De Oncologia | Urologia, Valencia
  - Hospital Universitario Y Politecnico La Fe | Oncologia Radioterapica, Valencia
- Sweden (2):
  - Goteborgs Universitet, Gothenburg
  - Skane University Hospital - Department of Urology, Malmo
- Taiwan (4):
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yet-Sen Cancer Centre, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- United Kingdom (5):
  - University College London Hospitals NHS Foundation Trust | University College Hospital (UCLH) - Cancer Clinical Trials Unit, London, Greater London
  - The Royal Marsden NHS Foundation Trust | The Royal Marsden Hospital - The Royal Marsden Clinical Trials Unit (CTU), London, Greater London
  - Imperial College Healthcare NHS Trust | Charing Cross Hospital - Cancer Services, London, Greater London
  - East and North Hertfordshire NHS Trust - Mount Vernon Hospital - Mount Vernon Cancer Centre (MVCC), Northwood, Middlesex
  - Royal Surrey NHS Foundation Trust | Royal Surrey County Hospital - Cancer Centre, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Morgans AK, Chehrazi-Raffle A, Niazi T, Shore ND, Ross AE, Roder A, Gomes AJ, Supiot S, Barthelemy P, Hatano K, Ruiz CBC, Yoshida S, Herrera-Imbroda B, Gratton M, Gschwend JE, Hope TA, Joensuu H, Kuss I, Le Berre MA, Dimova-Dobreva M, Fizazi K. Darolutamide plus androgen-deprivation therapy in high-risk biochemical recurrence of prostate cancer (ARASTEP). Future Oncol. 2025 Nov;21(27):3491-3498. doi: 10.1080/14796694.2025.2577633. Epub 2025 Nov 11. PMID 41216639
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/